CLINICAL TRIAL: NCT00716521
Title: Subject- And Investigator-Blinded, Sponsor-Open, Randomized, Single-Dose, Placebo-Controlled, 3-Way Crossover Study To Study Effect Of Treatment With Oral Zolpidem On Polysomnography And Actigraphy Measures In Healthy Volunteers
Brief Title: Effect Of Treatment With Oral Zolpidem On Polysomnography And Actigraphy Measures In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: A9001390
Record Dates: First submitted 2008-06-23; First posted 2008-07-16 (Estimated); Last update posted 2009-04-24 (Estimated); Status verified 2009-04

CONDITIONS: Methodology Study
Keywords: mobile actigraphy inpatient polysomnography actigraphy ambien
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): groups of 3-4 subjects for overnight polysomnography assessments
  Interventions: Drug: placebo
- Low dose Zolpidem (Experimental)
  Interventions: Drug: zolpidem
- High dose zolpidem (Experimental)
  Interventions: Drug: zolpidem

INTERVENTIONS:
Drug: placebo — single oral dose placebo
  Arms: Placebo
Drug: zolpidem — single oral dose, 5 mg zolpidem
  Arms: Low dose Zolpidem
Drug: zolpidem — single oral dose, 10 mg zolpidem
  Arms: High dose zolpidem

SUMMARY:
This study will assess the feasibility of conducting sleep studies in a clinical research unit environment. In addition, the sensitivity of polysomnography and mobile actigraphy technologies will be compared for evaluating sleep stages and sleep architecture.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* BMI 18-30 kg/m2
* body weight > 50 kg

Exclusion Criteria:

* no history of sleep disorder
* no concurrent medications
* no alcohol use
* no medical issues
* no smoking

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
onset to persistent sleep | minutes

SECONDARY OUTCOMES:
awakenings after sleep onset | minutes

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001390&StudyName=Effect%20Of%20Treatment%20With%20Oral%20Zolpidem%20On%0APolysomnography%20And%20Actigraphy%20Measures%20In%20Healthy%0AVolunteers%0A